CLINICAL TRIAL: NCT01713504
Title: Identification of New Markers in the Hypereosinophilic Syndrome
Acronym: SHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008_29; 2009-A00314-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hypereosinophilic Syndrome
MeSH Terms: conditions — Hypereosinophilic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypereosinophilic syndrome unexplained (Experimental)
  Interventions: Biological: biologie sample
- Hypereosinophilic syndrome explained (Active Comparator)
  Interventions: Biological: biologie sample
- Normal rate of eosinophilic (Sham Comparator)
  Interventions: Biological: biologie sample

INTERVENTIONS:
Biological: biologie sample — comparison of biomarkers between HES, HE biomarkers data and control arms

SUMMARY:
The purpose is to characterize new hypereosinophilic syndrome biomarkers more informative and more accessible compared to those that we have already thanks to a proteomic approach. This will help the investigators to diagnose the this disease.

ELIGIBILITY:
Inclusion Criteria:

* dated and signed informed consent
* virale serology negative or negative result less than 6 months
* virale serology negative for HBV or vaccinated patient
* insured
* virale serology negative or negative result less than 6 months
* negative pregnancy test or female menopause for at least 1 year

Exclusion Criteria:

* subject enable adult, under guardianship or under protective measures of justice
* Refusal or inability to give informed consent
* The hypereosinophilic syndrome explained origin other than than atopy, bullous pemphigoid, the Churg-Strauss syndrome and DRESS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-06-29 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The aim is to characterize, through an approach immunoprotéomique, new HES biomarkers more informative and easier access than those currently available to us. These biomarkers will help to the diagnosis of HES, compared with other causes of eosinophilia. | one month after patient inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Prin, MD PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lefevre G, Copin MC, Roumier C, Aubert H, Avenel-Audran M, Grardel N, Poulain S, Staumont-Salle D, Seneschal J, Salles G, Ghomari K, Terriou L, Leclech C, Morati-Hafsaoui C, Morschhauser F, Lambotte O, Ackerman F, Trauet J, Geffroy S, Dumezy F, Capron M, Roche-Lestienne C, Taieb A, Hatron PY, Dubucquoi S, Hachulla E, Prin L, Labalette M, Launay D, Preudhomme C, Kahn JE; French Eosinophil Network. CD3-CD4+ lymphoid variant of hypereosinophilic syndrome: nodal and extranodal histopathological and immunophenotypic features of a peripheral indolent clonal T-cell lymphoproliferative disorder. Haematologica. 2015 Aug;100(8):1086-95. doi: 10.3324/haematol.2014.118042. Epub 2015 Feb 14. PMID 25682606